CLINICAL TRIAL: NCT07324525
Title: Oral Health and Dental Care in Palliative Medicine: A Survey Study Among Patients and Members of the German Society for Palliative Medicine
Brief Title: Oral Health in Palliative Care: A Survey Study
Acronym: OH-PAL
Status: Not yet recruiting | Type: Observational
Sponsor: University Medical Center Goettingen (Other)
Responsible Party: Principal Investigator, Felix Marschner, Senior Physician, University Medical Center Goettingen
Other Study IDs: 24/12/25
Record Dates: First submitted 2025-12-17; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Oral Health Care; Oral Health-Related Quality of Life; Palliative Care; Palliative Care, Patient Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients in palliative care: Patients receiving palliative care at the Department of Palliative Medicine of University Medical Center Göttingen
- Members of the German Society for Palliative Medicine: Members of the German Society for Palliative Medicine, including healthcare professionals involved in palliative care across various disciplines

SUMMARY:
Oral health problems such as xerostomia or oral infections are common in palliative care patients and can significantly impair quality of life. Adequate dental care may contribute substantially to symptom control and well-being; however, oral health and dental services are often insufficiently integrated into palliative care practice. In addition, little is known about the level of awareness, knowledge, and interprofessional collaboration regarding oral health among palliative care professionals.

This prospective, non-interventional survey study aims to assess the relevance of oral health in palliative care by surveying both palliative care patients and healthcare professionals who are members of the German Society for Palliative Medicine. The study investigates patients' oral health status, oral health-related quality of life, and access to dental care, as well as professionals' knowledge, attitudes, and current practices related to oral health and dental care in palliative settings. The findings are intended to identify existing gaps and inform strategies for improved integration of dental expertise into palliative care.

DETAILED DESCRIPTION:
Oral complaints are highly prevalent among patients receiving palliative care and are frequently caused or exacerbated by systemic diseases, cancer therapies, and medication-related side effects. Conditions such as xerostomia, oral candidiasis, mucositis, and pain can substantially affect nutrition, communication, comfort, and overall quality of life. Despite this high burden, oral health and dental care are often not systematically addressed in palliative care, and dental professionals are rarely integrated into interdisciplinary care structures.

To date, there is limited evidence regarding how oral health is perceived by palliative care patients, how dental care is organized and accessed in palliative settings, and how well palliative care professionals are informed about common oral health problems and their management. Furthermore, barriers and facilitators of interprofessional collaboration between palliative care teams and dental professionals remain insufficiently explored.

This prospective, non-interventional survey study aims to evaluate the role of oral health in palliative care from both patient and professional perspectives. Members of the German Society for Palliative Medicine (DGP) will be invited to participate in an anonymous online survey distributed via email and newsletter, with reminders sent after six and twelve weeks. The questionnaire for healthcare professionals assesses the relevance of oral health and dental care in daily clinical practice, knowledge of common oral conditions such as xerostomia and candidiasis, use of information sources and continuing education, and the integration of oral health topics into professional training and education.

Palliative care patients will be recruited through direct personal approach and will complete a pseudonymized paper-based questionnaire. Patient-reported outcomes include current oral health status, presence of oral complaints, access to dental care, and oral health-related quality of life measured using the German version of the Oral Health Impact Profile 14.

As this is a survey-based study, no clinical examinations or interventions are performed. Participation consists solely of completing the questionnaire once and is not part of routine clinical care. Eligible participants include adult, consent-capable palliative care patients whose health status allows questionnaire completion, as well as consent-capable DGP members. Individuals under 18 years of age or unable or unwilling to provide informed consent are excluded.

Data collection is conducted at the University Medical Center Göttingen. The results are expected to provide insights into current deficits, educational needs, and structural challenges and to support the development of strategies for better integration of oral health and dental care into palliative care services.

ELIGIBILITY:
Inclusion Criteria:

* consent-capable patients receiving palliative care
* patients whose health status allows completion of a questionnaire
* consent-capable members of the German Society for Palliative Medicine

Exclusion Criteria:

* Participants under 18 years of age
* Individuals who are unable or unwilling to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population includes adult, consent-capable patients receiving palliative care at the Palliative Care Department of University Medical Center Göttingen, as well as consent-capable members of the German Society for Palliative Medicine (DGP). Patients are under the care of the palliative team at the clinic, and DGP members represent healthcare professionals involved in palliative care across various disciplines in Germany.
Sampling Method: Non-Probability Sample
Enrollment: 151 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
The prevalence (%) of oral mucositis among patients receiving palliative care | At baseline (single cross-sectional assessment)
The percentage (%) of German Society for Palliative Medicine members reporting insufficient knowledge regarding dental care in palliative settings. | At baseline (single cross-sectional assessment)

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center Goettingen, Göttingen, Germany, Germany

IPD SHARING:
Plan to Share IPD: No